CLINICAL TRIAL: NCT02652611
Title: The Effect of Sacroiliac (SI) Screw Removal on Patient-Reported Pain and Functional Outcomes After Open or Closed Reduction and Internal Fixation of Pelvic Fractures
Brief Title: Sacroiliac (SI) Screws: The Effect of SI Screw Removal on Patient-Reported Pain and Functional Outcomes
Acronym: SIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Marcus Sciadini, Associate Professor in Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00063838
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sacroiliac Joint; Pain; Pelvis
Keywords: Screw Removal vs. Non-screw removal; Complications; SI Screw Stabilization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Screw Removal (Experimental): Patients enrolled in the SI screw removal treatment group will undergo the surgery 5-9 months after the initial SI screw stabilization surgery. The surgeon will remove all screws that he/she is able and feels is appropriate for the patient. The patient will mobilize as per the surgeon's instructions and x-rays will be taken at follow-up clinic appointments as per standard of care to determine if the injury continues healing properly. If additional surgery is required or other complications arise, this will be recorded within the study follow-up forms.
  Interventions: Procedure: SI Screw Removal Surgery
- Non-screw Removal (Experimental): Patients enrolled in the Non-SI screw removal treatment group will not undergo surgical intervention to for removal of their SI screws. remove all screws that he/she is able and feels is appropriate for the patient. The patient will mobilize as per the surgeon's instructions and x-rays will be taken at follow-up clinic appointments as per standard of care to determine if the injury continues healing properly. If complications arise and/or the patient requires screw removal surgery, crossover will be allowed and recorded within study follow0up forms.
  Interventions: Procedure: Non-screw removal treatment (non-operative management)

INTERVENTIONS:
Procedure: SI Screw Removal Surgery
  Arms: Screw Removal
Procedure: Non-screw removal treatment (non-operative management)
  Arms: Non-screw Removal

SUMMARY:
Chronic pain following surgical stabilization of a pelvic fracture is very prominent and can have a major affect on a patient's quality of life. Persistent pain after radiographic evidence of fracture union commonly leads to implant removal. But, the routine removal of orthopaedic fixation devices after fracture healing remains an issue of debate.

DETAILED DESCRIPTION:
Many surgeons remember patients whose intractable, hardly explainable local symptoms and complaints of pain resolved quickly after a hardware-removal procedure. However, implant removal requires a second surgical procedure in scarred tissue, poses a risk for nerve damage, infection and re-fractures, and is not a guarantee of pain relief.

Rates of implant removal vary based on anatomic location and implant selection. Many studies have introduced and assessed the outcomes of hardware removal in the ankle, tibia and femur. But, there is currently no controlled trial that assesses the benefits and harms of sacroiliac (SI) screw removal in pelvic fracture patients.

Reports in literature are not consistent concerning the incidence of painful hardware and the outcome and pain relief after hardware removal. There is conflicting evidence that removing hardware decreases acute pain in ankle, tibia, and femur fractures but there is a need to explore the effect of SI screw removal in pelvic fracture patients. The investigators propose to prospectively randomize patients with a pelvic fracture requiring the use of SI screws for stabilization to removal versus non-removal of SI screws and track which group has less pain and need for narcotic pain medications.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 18 and 80 years of age, inclusive
* The patient has a pelvic fracture that required SI screw stabilization
* The patient has reached skeletal maturity
* The patient's pelvic fracture was the result of trauma (includes polytraumatized patients)
* The patient is English-speaking
* The patient's pelvic fracture was initially treated at Shock Trauma
* The patient is currently experiencing pain associated with his/her pelvic fracture
* The patient's surgeon agrees to randomization (the patient is amendable to either SI screw removal or non-screw removal treatment)
* The patient is able to be randomized between 4 and 8 months post-SI screw stabilization surgery at an orthopaedic follow-up appointment

Exclusion Criteria:

* The patient is non-ambulatory due to an associated spinal cord injury
* The patient was non-ambulatory pre-injury
* The patient is currently pregnant
* The patient is enrolled in another study that does not allow co-enrollment
* The patient is likely to have severe problems with maintaining follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Sciadini, MD, Principal Investigator — University of Maryland; Gerard Slobogean, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Shock Trauma Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobsen S, Honnens de Lichtenberg M, Jensen CM, Torholm C. Removal of internal fixation--the effect on patients' complaints: a study of 66 cases of removal of internal fixation after malleolar fractures. Foot Ankle Int. 1994 Apr;15(4):170-1. doi: 10.1177/107110079401500402. PMID 7951948
- [Background] Brown OL, Dirschl DR, Obremskey WT. Incidence of hardware-related pain and its effect on functional outcomes after open reduction and internal fixation of ankle fractures. J Orthop Trauma. 2001 May;15(4):271-4. doi: 10.1097/00005131-200105000-00006. PMID 11371792
- [Background] Dodenhoff RM, Dainton JN, Hutchins PM. Proximal thigh pain after femoral nailing. Causes and treatment. J Bone Joint Surg Br. 1997 Sep;79(5):738-41. doi: 10.1302/0301-620x.79b5.7345. PMID 9331026
- [Background] Keating JF, Orfaly R, O'Brien PJ. Knee pain after tibial nailing. J Orthop Trauma. 1997 Jan;11(1):10-3. doi: 10.1097/00005131-199701000-00004. PMID 8990026
- [Background] Court-Brown CM, Gustilo T, Shaw AD. Knee pain after intramedullary tibial nailing: its incidence, etiology, and outcome. J Orthop Trauma. 1997 Feb-Mar;11(2):103-5. doi: 10.1097/00005131-199702000-00006. PMID 9057144
- [Background] Busam ML, Esther RJ, Obremskey WT. Hardware removal: indications and expectations. J Am Acad Orthop Surg. 2006 Feb;14(2):113-20. doi: 10.5435/00124635-200602000-00006. PMID 16467186
- [Background] Gerbershagen HJ, Dagtekin O, Isenberg J, Martens N, Ozgur E, Krep H, Sabatowski R, Petzke F. Chronic pain and disability after pelvic and acetabular fractures--assessment with the Mainz Pain Staging System. J Trauma. 2010 Jul;69(1):128-36. doi: 10.1097/TA.0b013e3181bbd703. PMID 20093984
- [Background] Meyhoff CS, Thomsen CH, Rasmussen LS, Nielsen PR. High incidence of chronic pain following surgery for pelvic fracture. Clin J Pain. 2006 Feb;22(2):167-72. doi: 10.1097/01.ajp.0000174266.12831.a2. PMID 16428951
- [Background] Pohlemann T, Tscherne H, Baumgartel F, Egbers HJ, Euler E, Maurer F, Fell M, Mayr E, Quirini WW, Schlickewei W, Weinberg A. [Pelvic fractures: epidemiology, therapy and long-term outcome. Overview of the multicenter study of the Pelvis Study Group]. Unfallchirurg. 1996 Mar;99(3):160-7. German. PMID 8685720
- [Background] Hanson B, van der Werken C, Stengel D. Surgeons' beliefs and perceptions about removal of orthopaedic implants. BMC Musculoskelet Disord. 2008 May 24;9:73. doi: 10.1186/1471-2474-9-73. PMID 18501014
- [Background] Toms AD, Morgan-Jones RL, Spencer-Jones R. Intramedullary femoral nailing: removing the nail improves subjective outcome. Injury. 2002 Apr;33(3):247-9. doi: 10.1016/s0020-1383(01)00145-0. PMID 12084641
- [Background] Williams AA, Witten DM, Duester R, Chou LB. The benefits of implant removal from the foot and ankle. J Bone Joint Surg Am. 2012 Jul 18;94(14):1316-20. doi: 10.2106/JBJS.J.01756. PMID 22810403

RESULTS

PARTICIPANT FLOW:
Groups:
- Screw Removal: Patients enrolled in the SI screw removal treatment group will undergo the surgery 5-9 months after the initial SI screw stabilization surgery. The surgeon will remove all screws that he/she is able and feels is appropriate for the patient. The patient will mobilize as per the surgeon's instructions and x-rays will be taken at follow-up clinic appointments as per standard of care to determine if the injury continues healing properly. If additional surgery is required or other complications arise, this will be recorded within the study follow-up forms.
  SI Screw Removal Surgery
- Non-screw Removal: Patients enrolled in the Non-SI screw removal treatment group will not undergo surgical intervention to for removal of their SI screws. The patient will mobilize as per the surgeon's instructions and x-rays will be taken at follow-up clinic appointments as per standard of care to determine if the injury continues healing properly. If complications arise and/or the patient requires screw removal surgery, crossover will be allowed and recorded within study follow up forms.
  Non-screw removal treatment (non-operative management)
Period: Overall Study
Arm/Group | Screw Removal | Non-screw Removal
Started | 15 | 45
Completed | 14 | 14
Not Completed | 1 | 31

BASELINE CHARACTERISTICS:
Population: Based on the limited enrollment in the trial and the high rate of treatment crossover in the trial, we pooled the randomized trial and observational patients for this analysis. To mitigate this bias, we matched patients who underwent iliosacral screw removal to a control group of patients who retained their iliosacral screws.
Groups:
- Non-screw Removal: Patients enrolled in the Non-SI screw removal treatment group will not undergo surgical intervention to for removal of their SI screws. The patient will mobilize as per the surgeon's instructions and x-rays will be taken at follow-up clinic appointments as per standard of care to determine if the injury continues healing properly. If complications arise and/or the patient requires screw removal surgery, crossover will be allowed and recorded within study follow-up forms.
  Non-screw removal treatment (non-operative management)
- Total: Total of all reporting groups
Arm/Group | Screw Removal | Non-screw Removal | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Based on the limited enrollment in the trial and the high rate of treatment crossover in the trial, we pooled the randomized trial and observational patients for this analysis. To mitigate this bias, we matched patients who underwent iliosacral screw removal to a control group of patients who retained their iliosacral screws.
  years | 44 (16) | 34 (13) | 39 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 8 | 11 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 54
fracture classification [Count of Participants; unit: Participants] — APC I injuries show less than 2.5 cm of symphyseal widening and have no posterior instability APC II injuries show widening of the symphysis pubis and instability of the posterior pelvis APC III injuries are those associated with complete posterior ligamentous disruption.
  LC I injuries result from a lateral force delivered over the posterior aspect of the pelvis LC II injuries result from a more anteriorly directed force. LC III injuries result from greater force.
  Participants
    Anterior Posterior Compression 1 (APC1) | 0 | 1 | 1
    Anterior Posterior Compression 2 (APC 2) | 1 | 3 | 4
    Anterior Posterior Compression 3 (APC 3) | 1 | 3 | 4
    Lateral Compression 1 (LC 1) | 9 | 4 | 13
    Lateral Compression 2 (LC 2) | 3 | 1 | 4
    Lateral Compression 3 (LC 3) | 0 | 2 | 2
Area Deprivation Index [Mean (Standard Deviation); unit: units on a scale] — Socioeconomic status were measured using Area Deprivation Index (ADI). ADI is a mapping tool that displays the relative socioeconomic conditions of neighborhoods created from publicly-available data in the theoretical domains of income, education, employment and housing quality. ADIs are national percentile rankings from a low of 1 to a high of 100. A ranking of 1 indicates the lowest level of "disadvantage" within the nation and a ranking of 100 indicates the highest level of "disadvantage".
  units on a scale | 40 (18) | 49 (27) | 44.5 (22.5)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Within 6 Months After Iliosacral Screw Removal Using the Brief Pain Inventory (BPI)
Description: The BPI is presented on a 0-10 level visual analog scale with a 24-hour recall period. A level of 0 is described to the patients as "no pain," and "10" described as "pain as bad as you can imagine." The BPI includes four items: the worst pain the patient has felt in the last 24 hours, the least pain the patient has felt in the last 24 hours, the average pain the patient has felt in the last 24 hours, and the pain the patient feels right now. The BPI score is the average of the four items.
Time Frame: Up to 24 months post initial SI screw stabilization
Population: The study included patients aged 18-80 years with an unstable posterior pelvic ring fracture who underwent open or closed reduction and internal fixation with iliosacral screws. For inclusion, patients were screened for postoperative pain at a clinic visit between 4 and 8 months after their initial surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Non-screw Removal: Patients enrolled in the Non-SI screw removal treatment group will not undergo surgical intervention to for removal of their SI screws. The patient will mobilize as per the surgeon's instructions and x-rays will be taken at follow-up clinic appointments as per standard of care to determine if the injury continues healing properly. If complications arise and/or the patient requires screw removal surgery, crossover will be allowed and recorded within study follow0up forms.
  Non-screw removal treatment (non-operative management)
Arm/Group | Screw Removal | Non-screw Removal
Number analyzed (Participants) | 14 | 14
units on a scale | 3.7 (2.7) | 4.7 (3.0)
Statistical Analysis 1: Comparison: Screw Removal vs Non-screw Removal; We reported the average pain and function from 6 to 24 months postinjury with 95% confidence intervals (CIs) and summarized pain and function at 6, 9, 12, 18, and 24 months postinjury with means and standard deviations and medians with interquartile ranges; Test type: Superiority; p = 0.57, t-test, 2 sided; Odds Ratio (OR) = 0.3, 95% CI 2-sided [-0.8 to 1.4]

2. Secondary Outcome: Pelvic Function Within 6 Months After Iliosacral Screw Removal, Measured Using the Majeed Pelvic Outcome Score.
Description: The Majeed Pelvic Outcome Score is a clinically validated tool that assesses pain, working status, walking distance, sitting, sexual intercourse, walking aids, unaided gait, and walking distance. The score is reported on a 0-100 point scale with higher values indicating better pelvic function.
Time Frame: Up to 24 months post initial SI screw stabilization
Population: The study included patients aged 18-80 years with an unstable posterior pelvic ring fracture who underwent open or closed reduction and internal fixation with iliosacral screws.
Measure: Mean (Standard Deviation); unit: score on a scale of 0-100
Arm/Group | Screw Removal | Non-screw Removal
Number analyzed (Participants) | 14 | 14
score on a scale of 0-100 | 68.3 (17.8) | 63.6 (23.6)
Statistical Analysis 1: Comparison: Screw Removal vs Non-screw Removal; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-2.9 to 12.3]

ADVERSE EVENTS:
Time Frame: 24 months following surgery and enrollment into study
Description: The definitions do not differ.
Arm/Group | Screw Removal | Non-screw Removal
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/14
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screw Removal (N=14) | Non-screw Removal (N=14)
Bacteremia (Infections and infestations) | 0 (0) | 1 (3) — Patient readmitted 3 months post SI screw stabilization due to fever, elevated C reactive protein, and elevated erythrocyte sedimentation rate. Diagnosed with Bacteremia. Resolved non-operatively (4 weeks Ancef).
Unplanned surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient presents to outpatient clinic with foot-drop 12 months post SI screw stabilization (deficit present since trauma resulting in study injury). In attempt to correct deficit, surgeon conducted a lower extremity nerve decompression surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT02652611/Prot_SAP_000.pdf